CLINICAL TRIAL: NCT03203161
Title: A Prospective Observational Cohort Study Collecting Coordinated Clinical, Epidemiological, and Behavioural Data to Assess Safety and Efficacy of Surgical Treatment in Adolescent Morbid Obese Patients
Brief Title: Registry on Obesity Surgery in Adolescents
Acronym: ROSA
Status: Not yet recruiting | Type: Observational
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: P2017/CHIR/ROSA
Record Dates: First submitted 2017-06-22; First posted 2017-06-29 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Morbid Obesity; Bariatric Surgery; Adolescent Obesity
MeSH Terms: conditions — Obesity, Morbid; Pediatric Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bariatric surgery — Roux-and-Y Gastric Bypass or Sleeve gastrectomy

SUMMARY:
While bariatric surgery is established as a safe and effective alternative with well-defined risks for severely obese adults, little has been published on its use in children.

There are many unresolved questions concerning the long-term metabolic and psychological consequences of bariatric surgery in adolescents, and the difference with the adult population. The appropriate timing for bariatric surgery in young people, and the predictors of success and safety still need to be determined.

The aim of this long-term prospective study is therefore to establish the safety and efficacy profile of surgical procedures and to clarify whether reductions in morbidity and mortality outweigh the risks of serious surgical complications and lifelong nutritional deficiencies.

DETAILED DESCRIPTION:
The investigators will conduct a prospective observational cohort design study to collect data during standard clinical care of adolescent bariatric patients (younger than 18 years) who were operated (RYGB or SG) for weight loss.

Medical, psychological, behavioral, fitness and social data will be collected by medical personnel guided by checklists and prepared questionnaires. All non-invasive and invasive examinations will be performed following the existing protocol of the multidisciplinary group at the hospital (no alteration of normal standard care). Data regarding family environment (birthdays, weight, length, medication, comorbidities, smoking and education of parents and siblings) will also be obtained from caregivers of the patients.

ELIGIBILITY:
Inclusion Criteria:

* BMI (or projected BMI) > 40 kg/m² (projected BMI = weight over the age- and gender-specific BMI z-score defined as severe obesity corresponding at a projected BMI of 40 at the age of 18y) OR
* BMI ((or projected BMI) > 35 kg/m² (projected BMI = weight over the age- and gender-specific BMI z-score defined as severe obesity corresponding at a projected BMI of 35 at the age of 18y) + 1 or more of the following obesity-related comorbid conditions: Obstructive Sleep Apnea Syndrome, Non-alcoholic steatohepatitis, type 2 diabetes, hypertension, benign intracranial hypertension.
* Minimum 6 months of organized weight loss attempts before surgery (multidisciplinary follow-up)
* Completed most of their linear growth (Tanner stage ≥ IV, bone age ≥ 13 years in girls and ≥ 14 years in boys assessed by the Tanner and Whitehouse method)
* Capability and willingness to adhere to postoperative guidelines and prolonged surveillance
* Informed Consent Form (ICF) signed by patient and parents (or legal guardian)

Exclusion Criteria:

* psychological/psychiatric disorders that are decompensated or not efficiently treated
* severe and unstable eating disorders (e.g. binge-eating)
* signs of addictions or addictive behavior (alcohol or substance abuse)
* pregnancy or breastfeeding
* life-threatening multisystem organ failure
* uncontrolled or metastatic malignancy
* uncontrolled HIV infection
* hypercarbic respiratory failure
* active systemic infection or untreated endocrine dysfunction
* diseases threatening in the short term or lack of care (self-care or access to family or social support)
* medically correctable causes of obesity

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Resolution rate of baseline comorbidities associated with morbid obesity | 1 year after bariatric surgery
  comorbidities resolution rate will be expressed in %

SECONDARY OUTCOMES:
Resolution rate in baseline comorbidities associated with morbid obesity | 5 years after bariatric surgery
  comorbidities resolution rate will be expressed in %
Incidence of treatment-emergent adverse event | 30 days after bariatric surgery
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Incidence of treatment-emergent adverse event | 1 year after bariatric surgery
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Incidence of treatment-emergent adverse event | 5 years after bariatric surgery
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Overall mortality rate | 30 days after bariatric surgery
  Overall mortality rate will be expressed in %
Overall mortality rate | 1 year after bariatric surgery
  Overall mortality rate will be expressed in %
Overall mortality rate | 5 years after bariatric surgery
  Overall mortality rate will be expressed in %
Change from baseline in vitamin deficiencies | 1 year after bariatric surgery
  Change in vitamin deficiencies will be expressed in %
Change from baseline in vitamin deficiencies | 5 years after bariatric surgery
  Change in vitamin deficiencies will be expressed in %
Change from baseline in mineral deficiencies | 1 year after bariatric surgery
  Change in mineral deficiencies will be expressed in %
Change from baseline in mineral deficiencies | 5 years after bariatric surgery
  Change in mineral deficiencies will be expressed in %
Weight loss | 1 year after bariatric surgery
  weight loss will be reported in kg
Weight loss | 5 years after bariatric surgery
  weight loss will be reported in kg
Reduction in BMI | 1 year after bariatric surgery
  BMI will be reported in kg/m^2
Reduction in BMI | 5 years after bariatric surgery
  BMI will be reported in kg/m^2
Change from baseline in body mass composition | 2 years after bariatric surgery
  Change in Fat Mass and Lean Body Mass will be reported in kg
Change from baseline in body mass composition | 5 years after bariatric surgery
  Change in Fat Mass and Lean Body Mass will be reported in kg
Change from baseline in Eating behaviors after bariatric surgery | 1 year after bariatric surgery
  Change in Eating Behaviors behaviors will be assessed by Dutch Eating Behaviour Questionnaire (DEBQ) and will be reported in units on a scale
Change from baseline in Eating behaviors after bariatric surgery | 2 years after bariatric surgery
  Change in Eating Behaviors behaviors will be assessed by DEBQ questionnaire and will be reported in units on a scale
Change from baseline in Eating behaviors after bariatric surgery | 5 years after bariatric surgery
  Change in Eating Behaviors behaviors will be assessed by DEBQ questionnaire and will be reported in units on a scale
Change from baseline in quality of life after bariatric surgery | 1 year after bariatric surgery
  Change in Quality of Life will be assessed by PedsQL questionnaire and will be reported in units on a scale
Change from baseline in quality of life after bariatric surgery | 2 years after bariatric surgery
  Change in Quality of Life will be assessed by PedsQL questionnaire and will be reported in units on a scale
Change from baseline in quality of life after bariatric surgery | 5 years after bariatric surgery
  Change in Quality of Life will be assessed by PedsQL questionnaire (units on a scale)

CONTACTS AND LOCATIONS:
Overall Officials: Henri Steyaert, MD-PhD, Principal Investigator — Hôpital Universitaire Des Enfants Reine Fabiola (HUDERF)
Locations (3):
- Belgium (3):
  - CHU Saint Pierre, Brussels
  - Hôpital Universitaire Des Enfants Reine Fabiola, Brussels
  - Universitair Ziekenhuis Brussel (UZB), Brussels

IPD SHARING:
Plan to Share IPD: No